CLINICAL TRIAL: NCT05680402
Title: Effects of Soft Tissue Mobilization Technique and Piriformis Muscle Stretching Among Patients Having Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: Physiotherapy Clinic Iqra University Islamabad (Chak Shahzad) (Unknown); Noor Hospital Tarnol, Islamabad (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 339
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Clinical Trial in which group 1 will be of experimental group and group 2 will be of control group
Who Masked: Participant
Masking Description: Single Blind RCT in which only participants will not know about the type of treatment undergoing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Soft tissue mobilization
  Interventions: Other: Soft Tissue mobilization
- Group 2 (Active Comparator): Piriformis Stretching
  Interventions: Other: Piriformis Syndrome (Piriformis muscle stretching)

INTERVENTIONS:
Other: Soft Tissue mobilization — mobilization of soft tissues of body
  Arms: Group 1
Other: Piriformis Syndrome (Piriformis muscle stretching) — Stretching of Piriformis muscle
  Arms: Group 2

SUMMARY:
It is a randomized control trail in which soft tissue mobilization and piriformis stretching will be compared and study duration will be of five months

DETAILED DESCRIPTION:
Piriformis syndrome is one of the misdiagnosed syndromes and there is no evidence available for the proper diagnosis of this syndrome. Several interventions have been adopted in the clinical setting for improvement of piriformis syndrome including therapeutic ultrasound, myofascial release, stretching, dry needling, strengthening exercises of hip muscles and activity modification. There are several treatments available for this syndrome but no comparison studies have been reported yet on soft tissue mobilization and piriformis muscle stretching. The purpose for conducting this research is to assist in establishing the effectiveness of soft tissue mobilization technique and piriformis muscle stretching in piriformis syndrome by comparison between two abovementioned treatments

ELIGIBILITY:
Inclusion Criteria:

* Males and females with age between 25 and 45 years
* Patients with positive piriformis test
* Pain at least 3 according to numeric pain rating scale (NPRS)

Exclusion Criteria:

* History of hip pain due to any diagnosed hip pathology
* Leg length discrepancy
* Past history of spinal surgery
* Spinal tuberculosis
* Rheumatoid disease,

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 1 week
  Zero means non pain and 10 Means worst type of pain
Modified Oswestry Disability Index (ODI) questionnaire | 1 Week
  A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kamran, M.Phil*, Principal Investigator — Al Nafees medical College Hospital
Locations (1):
- Physiotherapy Clinic Iqra University Islamabad (Chak Shahzad), Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No
Have not decided yet